CLINICAL TRIAL: NCT04529512
Title: INtravitreal and Aqueous Dexamethasone Levels After DEXtenza
Acronym: INDEX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nathan Steinle (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nathan Steinle, Principal Investigator, California Retina Consultants
Organization: California Retina Consultants (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INDEX
Record Dates: First submitted 2020-08-11; First posted 2020-08-27 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Ocular Disease Requiring Surgery
MeSH Terms: interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Receiving DEXTENZA® 1-3 days prior to surgery (Experimental): Participants to receive DEXTENZA® 1-3 days prior to surgery
  Interventions: Drug: DEXTENZA®
- Receiving DEXTENZA® 1-2 weeks prior to surgery (Experimental): Participants to receive DEXTENZA® 1-2 weeks prior to surgery
  Interventions: Drug: DEXTENZA®
- Receiving DEXTENZA® 1 month prior to surgery (Experimental): Participants to receive DEXTENZA® 1 month prior to surgery
  Interventions: Drug: DEXTENZA®
- Not receiving the DEXTENZA® implant (No Intervention): Participants will not receive the DEXTENZA® implant

INTERVENTIONS:
Drug: DEXTENZA® — DEXTENZA® is a corticosteroid implant indicated for the treatment of ocular pain following ophthalmic surgery. DEXTENZA® is inserted into the lower lacrimal punctum into the canaliculus by the physician following ophthalmic surgery. A single DEXTENZA® releases a 0.4 mg dose of dexamethasone for up to 30 days following insertion. DEXTENZA® is preservative free, resorbable and does not require removal. Saline irrigation or manual expression can be performed to remove the insert, if necessary.
  Other Names: dexamethasone ophthalmic insert 0.4mg
  Arms: Receiving DEXTENZA® 1 month prior to surgery; Receiving DEXTENZA® 1-2 weeks prior to surgery; Receiving DEXTENZA® 1-3 days prior to surgery

SUMMARY:
A prospective, open-label, interventional study to determine intraocular concentration levels of dexamethasone following use of the DEXTENZA® implant.

DETAILED DESCRIPTION:
On December 3rd, 2018, DEXTENZA® was approved by the FDA for the treatment of ocular pain following ophthalmic surgery. On June 21st, 2019, the FDA approved a Supplemental New Drug Application (sNDA) for DEXTENZA® to include the treatment of ocular inflammation following ophthalmic surgery as an additional indication.

DEXTENZA® is a corticosteroid implant indicated for the treatment of ocular pain following ophthalmic surgery. DEXTENZA® is inserted into the lower lacrimal punctum into the canaliculus by the physician following ophthalmic surgery. A single DEXTENZA® releases a 0.4 mg dose of dexamethasone for up to 30 days following insertion. DEXTENZA® is preservative free, resorbable and does not require removal. Saline irrigation or manual expression can be performed to remove the insert, if necessary.

In the two phase III trials, patients were given DEXTENZA® or its vehicle immediately after cataract surgery. In the first study, 80 percent of DEXTENZA®-treated patients (n=164) were pain-free at the eighth day compared to 43 percent of vehicle-treated patients (n=83) (p<0.0001). In the second trial, 77 percent of patients on active drug (n=161) were pain-free at the eighth day vs. 59 percent of those on the vehicle.1

Safety was assessed from the three Phase 3 clinical trials and a Phase 2 clinical trial.1,2 Overall, 567 subjects were exposed to DEXTENZA®. The most common ocular adverse reactions in subjects treated with DEXTENZA® were: anterior chamber inflammation including iritis and iridocyclitis (10%), increased intraocular pressure (6%), reduced visual acuity (2%), cystoid macular edema (1%), corneal edema (1%), eye pain (1%), and conjunctival hyperemia (1%). The most common non-ocular adverse event was headache (1%).

Though DEXTENZA has been found to be safe and effective, it is a relatively new therapy and a randomized prospective study looking at dexamethasone and pain levels following retinal surgery has not yet been done. The purpose of this study is to provide real-world intraocular dexamethasone concentration levels in subjects implanted with DEXTENZA as well as to confirm the reduction of pain in patients undergoing retinal surgery is the same as subjects who underwent cataract surgery in the phase III studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of California Retina Consultants undergoing vitrectomy surgery
2. Must be 18 years old or older
3. Must be able to provide consent

Exclusion Criteria:

1. Must not have been treated with DEXTENZA® prior to joining the study.
2. May not have more than one DEXTENZA® implant.
3. May not be currently using an dexamethasone product during the course of the study or within 4 weeks prior to enrolling in the study.
4. Subject has active corneal, conjunctival or canalicular infections, including:

   i. Epithelial herpes simplex keratitis (dendritic keratitis)

   ii. Vaccini

   iii. Varicella

   iv. Mycobacterial infections

   v. Fungal diseases of the eye

   vi. Dacryocystitis
5. Any abnormal lid or punctum anatomy that would preclude or make inappropriate the placement of the insert (e.g., severe ectropion or punctal stenosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Intraocular dexamethasone levels | 8 months
  The primary objective is to determine intraocular dexamethasone levels by obtaining aqueous and intravitreal samples at the time of routine retina surgery after placement of DEXTENZA® prior to surgery; tear films will also be analyzed for osmolarity and dexamethasone levels.prior to starting the vitrectomy procedure (including eye prep), the physician will collect the subject's tear film for assessment of osmolarity and dexamethasone levels using a Schirmer test strip which will be stored in an Eppendorf tube on ice until it can be frozen and shipped to a lab for analysis.

SECONDARY OUTCOMES:
Post-operative pain levels | 8 months
  The secondary objective of this study is to assess post-operative pain levels in subjects with or without the DEXTENZA® implant following retinal surgery. This will be assessed using a pain post-surgery questionnaire.This will be assessed using a pain post-surgery questionnaire consisting of an an 11-point likert scale (0-10), with 0 being no pain and 10 being excruciating pain

CONTACTS AND LOCATIONS:
Overall Officials: Gabe Gordon, PhD, Study Director — Director of Research; Nathan Steinle, MD, Principal Investigator — Physician
Locations (3):
- United States (3):
  - California Retina Consultants, Paso Robles, California
  - California Retina Consultants, San Luis Obispo, California
  - California Retina Consultants, Santa Maria, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be published in a peer-review journal once the study is completed.
Time Frame: Don't know yet
Access Criteria: Don't know yet

REFERENCES:
- [Background] Tyson SL, Bafna S, Gira JP, Goldberg DF, Jones JJ, Jones MP, Kim JK, Martel JM, Nordlund ML, Piovanetti-Perez IK, Singh IP, Metzinger JL, Mulani D, Sane S, Talamo JH, Goldstein MH; Dextenza Study Group. Multicenter randomized phase 3 study of a sustained-release intracanalicular dexamethasone insert for treatment of ocular inflammation and pain after cataract surgery. J Cataract Refract Surg. 2019 Feb;45(2):204-212. doi: 10.1016/j.jcrs.2018.09.023. Epub 2018 Oct 24. PMID 30367938
- [Background] Torkildsen G, Abelson MB, Gomes PJ, McLaurin E, Potts SL, Mah FS. Vehicle-Controlled, Phase 2 Clinical Trial of a Sustained-Release Dexamethasone Intracanalicular Insert in a Chronic Allergen Challenge Model. J Ocul Pharmacol Ther. 2017 Mar;33(2):79-90. doi: 10.1089/jop.2016.0154. Epub 2017 Jan 10. PMID 28072552